CLINICAL TRIAL: NCT05629728
Title: Effect of Tai Chi on Physical and Cognitive Function Among Frail Older Adults
Brief Title: Tai Chi for Improving Functions of Frail Older Adults
Acronym: AAproject
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chungnam National University (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Rhayun Song, Professor, Chungnam National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ChungnamNU4
Record Dates: First submitted 2022-11-12; First posted 2022-11-29 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Frailty
Keywords: Tai Chi; frail; older adults
MeSH Terms: conditions — Frailty | interventions — Aquatic Therapy

STUDY DESIGN:
Intervention Model Description: the frail older adults recruited from the community, randomly assigned to either the experimental group or the wait-list control group.
Who Masked: Outcomes Assessor
Masking Description: the assessor will be blinded for the group assignment. trained research assistant will conduct the pretest and posttest measures, not involved in providing the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- frail elderly-TC (Experimental): Tai Chi group received 12 weeks of Tai Chi exercise program with 12 week follow-up, twice a week, 60 min per session led by a trained Tai Chi instructor
  Interventions: Behavioral: Tai Chi exercise
- frail elderly-WC (No Intervention): control group received no intervention for 12 weeks, and will be provided the chance to participate in Tai Chi program if they choose.

INTERVENTIONS:
Behavioral: Tai Chi exercise — Sun-style Tai Chi (21 forms)
  Arms: frail elderly-TC

SUMMARY:
The goals of this study are to examine the physical function, cognitive function, and quality of life among frail elderly residing in the community

DETAILED DESCRIPTION:
This randomized clinical trial recruited 100 frail older adults, assigned to either the Tai Chi group or the wait-list control group. Tai Chi intervention will be provided to the Tai Chi group for 12 weeks with 12-week follow-up and pretest and posttest measures will be conducted.

The primary outcome is the function variables (physical function of balance, flexibility, mobility; cognitive function of MOCA-K) The secondary outcome is quality of life measured by SF12.

ELIGIBILITY:
Inclusion Criteria:

* being frail (3 out of the following 5 criteria): feeling fatigued, difficulty climbing 10 stairs without help, difficulty walking 300m without help, more than 5 chronic illness, weight loss 5 % or more past 1-5 years
* living in the community
* able to participate in Tai Chi program twice a week

Exclusion Criteria:

* participated in any formal exercise program past 6 months
* not have transportation to come to the class

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-28 (Estimated)

PRIMARY OUTCOMES:
physical function - balance | changes from pretest to 12 week posttest scores
  balance was assessed using a one-leg-standing balance test (OLST)
physical function - flexibility | changes from pretest to 12 week posttest scores
  flexibility was assessed by the standard sit-and-reach test (SSRT)
physical function - mobility | changes from pretest to 12 week posttest scores
  mobility was assessed by the Timed Up and Go test (TUG)
cognitive function | changes from pretest to 12 week posttest scores
  MOCA-K (Korean version of Montreal Cognitive Assessment) was used with the maximum score of 30. (more than 23 is normal and less than 13 is dementia, more cognitively impaired)

SECONDARY OUTCOMES:
Short Form health survey 12 (SF12) | changes from pretest to 12 week posttest scores
  Short Form health survey 12 which consists of eight dimensions: general health, physical functioning, role physical, body pain, vitality, social functioning, role emotional, and mental health. two summary scores for the physical and mental components of health-related QoL are calculated by using the weighted means for the eight domains. Higher scores indicate better health-related QoL.

CONTACTS AND LOCATIONS:
Overall Officials: Rhayun Song, PhD, Principal Investigator — Chungnam National University
Locations (1):
- Chungnam National University, Daejeon, South Korea

IPD SHARING:
Plan to Share IPD: Yes
unidentified data or study protocol can be shared at the completion of publication
Supporting Information: Study Protocol, CSR
Time Frame: December, 2025
Access Criteria: researchers or reviewers with request